CLINICAL TRIAL: NCT03850522
Title: Phase IIa Trial of PD-L1 Peptide Vaccination as Monotherapy in High Risk Smoldering Multiple Myeloma
Brief Title: PD-L1 Peptide Vaccination in High Risk Smoldering Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient recruitment within planned enrolmentperiod.
Sponsor: Lene Meldgaard Knudsen (Other)
Collaborators: IO Biotech (Industry)
Responsible Party: Sponsor-Investigator, Lene Meldgaard Knudsen, Head of Department, Department of Hematology, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MY18H2; 2018-003990-93 (EudraCT Number)
Record Dates: First submitted 2019-02-19; First posted 2019-02-21 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Smoldering Multiple Myeloma
Keywords: smoldering; myeloma; vaccination; PD-L1; high-risk
MeSH Terms: conditions — Smoldering Multiple Myeloma; Neoplasms, Plasma Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vaccination (Experimental): Vaccination with PD-L1 peptide
  Interventions: Biological: PD-L1 peptide

INTERVENTIONS:
Biological: PD-L1 peptide — PD-L1 peptide (100 micrograms) emulsified with the adjuvant Montanide ISA-51 given subcutaneously 10 times every second week over the course of 26 weeks including a five-week break.
  Other Names: IO103

SUMMARY:
This study is evaluating a new vaccine against PD-L1 as a possible treatment for high-risk smoldering multiple myeloma.

DETAILED DESCRIPTION:
Smoldering multiple myeloma is an asymptomatic disorder with an annual risk of 10% of progression to the incurable cancer multiple myeloma. While many patients live for many years without progression, high risk patients have a median risk of progression of 29 months. No therapy has been approved for this indication. New treatments with limited adverse events are in high demand for this unmet medical need. An effective peptide vaccine would represent an ideal candidate, since vaccines generally have very low levels of side effects.

This study will explore if vaccination against the immune checkpoint molecule PD-L1 leads to responses in patients with high risk smoldering myeloma. PD-L1 is thought to play a role in the rate of progression from smoldering myeloma to symptomatic myeloma. Targeting this pathway with little risk of adverse events would potentially prevent or delay progression to symptomatic myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Patient has confirmed SMM according to a definition derived from the International Myeloma Working Group (IMWG) definition (International Working Group, 2003)

  1. Serum M-component >30g/L and/or
  2. Urine M-component ≥ 500mg/24 hours and/or
  3. ≥10% clonal plasma cells in bone marrow
  4. and no CRAB criteria or myeloma defining events (see exclusion criteria)
* High risk of progression to symptomatic multiple myeloma defined by the presence of ≥ 2 of the risk factors below:

  * Bone marrow Plasma Cells (BMPCs) ≥ 20%
  * M-component > 2g/dL
  * FLC ratio > 20
* Age ≥18 years
* Performance status ≤ 2 (ECOG-scale)
* Expected survival > 3 months
* Sufficient liver function, i.e.

  1. ALAT < 2.5 upper normal limit, i.e. ALAT <112 U/l
  2. Bilirubin < 30 U/l
* Women agreement to use contraceptive methods with a failure rate of < 1% per year during the treatment period and for at least 120 days after the last treatment.
* For men: agreement to use contraceptive measures and agreement to refrain from donating sperm.
* The accepted contraceptive methods are

  * Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation. Oral, intravaginal or transdermal.
  * Progestogen-only hormonal contraception associated with inhibition of ovulation. Oral, injectable, implantable.
  * Intrauterine device (IUD)
  * Intrauterine hormone-releasing system (IUS)
  * Bilateral tubal occlusion
  * Vasectomized partner
  * Sexual abstinence

Exclusion Criteria:

* Non-secretory myeloma
* Patients fulfilling CRAB criteria:

  i. C: Hypercalcemia,

  1. s-Ca-ion >1,40 mmol/L, attributable to myeloma ii. R: Renal failure
  1. Estimated or measured creatinine clearance <40ml/min, attributable to myeloma
  2. Increased s-creatinine, attributable to myeloma
  3. Decrease in estimated or measured creatinine clearance <35% within a year, attributable to myeloma
  4. Renal biopsy-verified renal changes attributable to myeloma iii. A: Anemia, Hgb < 6,3mmol/L (10g/dl), attributable to myeloma iv. B: Bone lesions on X-ray, CT or PET-CT
* Evidence of myeloma defining events i. Clonal bone marrow plasma cell percentage ≥ 60% ii. Ratio of involved/uninvolved serum free light chain ratio ≥ 100 iii. >1 focal lesions on MRI studies, if clinically indicated
* Plasma cell leukemia
* Signs of amyloidosis
* Other malignancies in the medical history excluding basal cell carcinoma of the skin, squamous cell carcinoma of the skin or in situ cervical cancer and patients cured for another malignant disease with no sign of relapse two years after ended treatment.
* Significant medical condition per investigators judgement e.g. severe Asthma/COPD, poorly regulated heart condition, insulin dependent diabetes mellitus.
* Acute or chronic viral infection e.g. HIV, hepatitis or tuberculosis
* Serious known allergies or earlier anaphylactic reactions.
* Known sensibility towards Montanide ISA-51
* Any active autoimmune diseases e.g. autoimmune neutropenia, thrombocytopenia or hemolytic anemia, systemic lupus erythematosus, scleroderma, myasthenia gravis, autoimmune glomerulonephritis, autoimmune adrenal deficiency, autoimmune thyroiditis etc.
* Pregnant and breastfeeding women.
* Fertile women not using secure contraception with a failure rate less than < 1%
* Patients taking immune suppressive medications incl. corticosteroids and methotrexate at the time of enrollment
* Psychiatric disorders that per investigator judgment could influence compliance.
* Treatment with other experimental drugs
* Concurrent treatment with other anti-cancer drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
Overall response rate | Planned analysis cut-off per patient: two weeks after last vaccination.
  Overall response rates (ORR) defined by IMWG criteria as PR+VGPR+CR+sCR during treatment and two weeks after end of treatment per patient.

SECONDARY OUTCOMES:
Immunogenicity of the PD-L1 vaccine | Samples taken before, during and two weeks after last vaccination.
  Blood, skin biopsies and bone marrow samples will be assessed with ELISPOT assays for levels of immune response to the vaccine.
Incidence of Treatment Emergent Adverse Events | Planned analysis cut-off per patient: two weeks after last vaccination
  Safety analysis will be conducted using the Safety Population defined as any patient receiving one dose of study treatment. For toxicity reporting, all adverse events and laboratory abnormalities will be graded and analyzed using CTCAE version 4 as appropriate.
Progression-free survival (PFS) | Planned analysis 2 years and 5 years post initiation of therapy.
  PFS from diagnosis is defined as the time from diagnosis to the disease progression or death from any cause. Patients who have not progressed or died are censored at the date last known progression-free. This will be compared with published progression rates.
Time to progression (TTP) | Planned analysis 2 years and 5 years post initiation of therapy.
  Time from diagnosis of SMM to progression to symptomatic myeloma compared to historical controls. Progression is defined as biochemical or diagnostic progression in accordance with the 2014 IMWG criteria for diagnosis of multiple myeloma which includes the classic CRAB-criteria as well as: Clonal bone marrow plasma cell percentage ≥ 60%, Free light chain ratio ≥ 100 (Involved FLC level must be ≥ 100mg/L),> 1 focal lesion on MRI studies (at least 5 mm in size)
Overall survival (OS) | Planned analysis 2 years and 5 years post initiation of therapy.
  OS from diagnosis is defined as the time from diagnosis to the death of the patient.

OTHER OUTCOMES:
Quality of Life (QoL) | Baseline and up to two weeks after last vaccination
  measured by change in European Organization for Research and Treatment of Cancer (EORTC) QLQ-30.
Quality of Life (QoL) | Baseline and up to two weeks after last vaccination
  measured by change in EuroQoL 5D-5-Level (EQ-5D-5L).
Quality of Life (QoL) | Baseline and up to two weeks after last vaccination
  measured by change in and Hospital Anxiety and Depression Scale (HADS).

CONTACTS AND LOCATIONS:
Overall Officials: Nicolai Jørgensen, MD, Principal Investigator — Department of Hematology
Locations (1):
- Department of Hematology, Universityhospital Herlev and Gentofte, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: Undecided